CLINICAL TRIAL: NCT02011308
Title: The Effect of KTP Green Light Prostatectomy (120W) Compared With TUR-P When Treating Benign Prostatic Hyperplasia (BPH), a Prospective Randomized Study
Brief Title: KTP (Potassium-titanyl-phosphate) Laser Versus TUR-P (Transurethral Resection of Prostate)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: University of Turku (Other); Tampere University (Other); South Ostrobothnia Health Care District (Other); Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Hannu Koistinen, Urologist, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34/13/03/02/08
Record Dates: First submitted 2012-02-21; First posted 2013-12-13 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: BPH (Benign Prostatic Hyperplasia)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Green Light Laser (Active Comparator)
  Interventions: Device: Green light Laser; Device: Transurethral Resection of the Prostate (TURP)
- TURP (Active Comparator): Transurethral Resection of the Prostate
  Interventions: Device: Green light Laser; Device: Transurethral Resection of the Prostate (TURP)

INTERVENTIONS:
Device: Green light Laser — Laser vs TURP
Device: Transurethral Resection of the Prostate (TURP) — Laser vs TURP

SUMMARY:
The purpose of this study is to compare safety and efficacy of Green Light PVP (Photoselective Vaporisation of the Prostate) compared to TUR-P.

ELIGIBILITY:
Inclusion Criteria:

* Men undergoing surgery for BPH

Exclusion Criteria:

* Previous prostate surgery
* Carcinoma of the prostate
* Neurogenic bladder
* Bladder carcinoma

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2011-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
IPSS (International Prostate Symptom Score) | 12 months
  symptom

SECONDARY OUTCOMES:
DAN-PSS (Danish Prostate Symptom Score) | 3, 6 and 12 months
  symptom
Maximum flow rate (Qmax) | 3, 6 and 12 months
Residual urine | 3, 6 and 12 months
Length of catheterization | Postoperative recovery
Length of hospital stay | Postoperative recovery
Perioperative bleeding | Time of operation
IIEF (International Index of Erectile Function questionnaire) | 12 months
  Erectile Dysfunction
TRUS (transrectal ultrasound) | 12 months
  Measurement of prostate size

CONTACTS AND LOCATIONS:
Overall Officials: Hannu T Koistinen, M.D., Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland